CLINICAL TRIAL: NCT06947538
Title: Adaptive Interventions to Improve Posttraumatic Stress Disorder (PTSD) Treatment Access, Engagement, and Effectiveness in Routine Care
Brief Title: Stepped Care for Posttraumatic Stress Disorder Study
Acronym: STEPPS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: H-45694; 1R01MH138549-01 (NIH)
Record Dates: First submitted 2025-04-21; First posted 2025-04-27 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Post Traumatic Stress Disorder
Keywords: Stepped Care; Skills training in affective and interpersonal regulation (STAIR); Digital Mental Health Intervention; Written Exposure Therapy (WET); Adaptive Interventions
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: This study uses a Sequential, Multiple Assignment, Randomized Trial (SMART) design. All participants enrolled will receive access to webSTAIR at baseline ("initial treatment").
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- webSTAIR, webSTAIR to WET (Active Comparator): First, offer skills-focused digital mental health intervention (DMHI); then switch to clinician-administered trauma-focused behavioral treatment for nonresponders and continue skills-focused DMHI for responders.
  Interventions: Behavioral: webSTAIR; Behavioral: Clinician administered WET
- webSTAIR+coaching, webSTAIR+coaching to WET (Active Comparator): First, offer skills-focused DMHI plus community health worker (CHW) coaching; then add clinician-administered trauma-focused behavioral treatment for nonresponders and continue skills-focused DMHI plus CHW coaching for responders.
  Interventions: Behavioral: WebSTAIR plus coaching; Behavioral: Clinician administered WET
- webSTAIR, webSTAIR to Brief STAIR (Active Comparator): First, offer skills-focused DMHI; then add clinician-administered skills-focused behavioral treatment for nonresponders and continue skills-focused DMHI for responders.
  Interventions: Behavioral: webSTAIR; Behavioral: Clinician administered Brief STAIR
- webSTAIR+coaching, websTAIR+coaching to Brief STAIR (Active Comparator): First, offer skills-focused DMHI plus CHW coaching; then add clinician-administered skills-focused behavioral treatment for nonresponders and continue skills-focused DMHI plus CHW coaching for responders.
  Interventions: Behavioral: WebSTAIR plus coaching; Behavioral: Clinician administered Brief STAIR

INTERVENTIONS:
Behavioral: webSTAIR — WebSTAIR consists of 10 online modules that provide psychoeducation on trauma and emotions and teach skills to improve coping with emotions and strengthen interpersonal relationships. Modules are completed at the participants' own pace and utilize interactive exercises, and audio and video components to aid in delivery.
  Arms: webSTAIR, webSTAIR to Brief STAIR; webSTAIR, webSTAIR to WET
Behavioral: WebSTAIR plus coaching — WebSTAIR with up to five 30-min coaching sessions with a CHW will focus on guiding participants through the program, discussing exercises that are valuable or problematic, and reviewing module content.
  Arms: webSTAIR+coaching, webSTAIR+coaching to WET; webSTAIR+coaching, websTAIR+coaching to Brief STAIR
Behavioral: Clinician administered Brief STAIR — Brief STAIR is a brief, low intensity, therapy that utilizes psychoeducation, coping skills training, and does not include recounting of the trauma memory, making it highly tolerable. It will be delivered by mental health clinicians in five to six 30-minute individual sessions.
  Arms: webSTAIR+coaching, websTAIR+coaching to Brief STAIR; webSTAIR, webSTAIR to Brief STAIR
Behavioral: Clinician administered WET — WET is a brief, high intensity, exposure-based treatment delivered by mental health clinicians consisting of six 30-minute individual sessions that cover treatment rationale, psychoeducation about PTSD, and directing participants to write in session about their traumatic experience using scripted instructions.
  Arms: webSTAIR+coaching, webSTAIR+coaching to WET; webSTAIR, webSTAIR to WET

SUMMARY:
Less than 20% of people with PTSD receive any treatment. This study extends a program of research by the investigator focused on developing adaptive (stepped) interventions for PTSD. The adaptive intervention sequences a digital mental health intervention (DMHI) and brief trauma- and skills-focused treatments for PTSD. The selected treatments are brief and scalable and less burdensome to systems of care. These treatments are: web-administered Skills Training in Affective and Interpersonal Regulation (webSTAIR), Brief STAIR, and Written Exposure Therapy (WET).

DETAILED DESCRIPTION:
This study uses a Sequential, Multiple Assignment, Randomized Trial (SMART) design. All participants enrolled will receive access to webSTAIR at baseline ("initial treatment").

Nonresponders at 4 weeks are randomized to either continue webSTAIR or webSTAIR plus community health worker coaching ("stage 1 treatments").

Nonresponders at 8 weeks are re-randomized to clinician-administered treatments, either Brief STAIR or WET ("stage 2 treatments").

Nonresponse is defined as less than a 15-point decrease in PTSD symptom severity, as measured by the PTSD Checklist for DSM-5 (PCL-5).

The objectives of this study are to:

* examine the main effects of stage 1 treatments, stage 2 treatments, and embedded
* adaptive interventions on PTSD symptom severity.
* confirm mechanisms of change established in the extant PTSD literature
* identify patient-level moderators of change in PTSD symptoms severity at 18 weeks

ELIGIBILITY:
Inclusion criteria:

Assessed at pre-screening

* Boston Medical Center primary care patient
* At least 18 years of age
* Access to computer or mobile device
* Able to receive treatments in English or Spanish
* Able to read at 4th grade level

Assessed at baseline

* Endorsement of Criterion A trauma using the Life Events Checklist for the DSM-5 (LEC-5), assessed at baseline
* PTSD diagnosis, confirmed by the Clinician-Administered PTSD Scale for the DSM-5 (CAPS-5) assessed at baseline
* Clinically appropriate for outpatient level of care
* Stable on psychotropic medication for >4 weeks

Exclusion criteria:

Assessed at pre-screening

• Patient is currently engaged in clinician-administered therapy

Assessed at baseline (clinician interview)

* Patient is not clinically appropriate for outpatient level of care.
* Acute risk for suicidal thoughts or behaviors, assessed by the Columbia Suicide Severity Rating Scale, administered by research clinician at baseline.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 428 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2029-06 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
PTSD symptom severity | baseline, 4 weeks, 8 weeks, 18 weeks, 30 weeks
  This outcome will be assessed by the PTSD Checklist for the DSM-5 (PCL-5), a 20-item self-report measure that evaluates the degree to which individuals have been bothered by PTSD symptoms in the past month tied to their most distressing event. Total scores ranging from 0 to 80, and a score of 31-33 or higher suggests probable PTSD and potential benefit from treatment.
Treatment retention | 4 weeks, 8 weeks, 18 weeks
  as the proportion (%) of participant who complete 60% of interventions in the treatment windows.
Treatment acceptability | 4 weeks, 8 weeks, 18 weeks, 30 weeks
  This outcome will be assessed with the Client Satisfaction Questionnaire 8 [CSQ-8], a 8-item instruction where scores are summed across items once. Items 2, 4, 5, and 8 are reverse scored. Total scores range from 8 to 32, with the higher number indicating greater satisfaction.

SECONDARY OUTCOMES:
Trauma coping | baseline, 4 weeks, 8 weeks, 18 weeks, 30 weeks
  This outcome will be assessed with the Trauma Coping Self-Efficacy Scale (TCSE, a 9-item instrument with items rated on a 7-point scale (1=not at all capable to 7=totally capable) and a total score calculated by averaging the item responses, Higher scores suggest better trauma coping.
Treatment expectancy | baseline, 4 weeks, 8 weeks, 18 weeks, 30 weeks
  This outcome will be assessed with the Treatment Expectancy Questionnaire (TEQ), is a multidimensional scale measuring participants' expectations of medical and psychological treatments, scored by adding up scores on each item to yield a total score, with higher scores indicating stronger expectations.
Mental health stigma | baseline, 4 weeks, 8 weeks, 18 weeks, 30 weeks
  This outcome will be assessed with the Consumer Experiences of Stigma Questionnaire (CESQ), using a 5-point Likert scale (never to very often) for each item, with higher scores indicating greater stigma experienced.
Medical mistrust | baseline, 4 weeks, 8 weeks, 18 weeks, 30 weeks
  This outcome will be assessed with the Group-Based Medical Mistrust Scale (GBMMS), a 12-item measure that assesses suspicion of mainstream health care systems and health care professionals and the treatment provided to individuals. The response key is a Likert-type scale ranging from 1 (strongly disagree) to 5 (strongly agree) and the score range is 12 to 60. Higher scores suggest more medical distrust.
Posttraumatic cognitions | baseline, 4 weeks, 8 weeks, 18 weeks, 30 weeks
  This outcome will be assessed with the 9-item brief version of the posttraumatic cognitions inventory (PTCI-9). It is scored by averaging the responses to its nine items (a Likert-type scale from 1 to 7) to get a total score ranging from 1 to 7. Higher scores reflect greater endorsement of negative posttraumatic cognitions.
Pathological fear extinction | baseline, 4 weeks, 8 weeks, 18 weeks, 30 weeks
  This outcome will be assessed with the subjective units of distress (SUDs), a simple self-assessment tool used to quantify the intensity of distress or anxiety an individual feels at a particular moment. Scores can range from 0 to 10 with a score of 0 indicating complete calmness, while 10 signifies the highest level of distress imaginable.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Valentine, PhD, Principal Investigator — Boston Medical Center, Psychiatry
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No